CLINICAL TRIAL: NCT03389139
Title: Comparison of the Effects of Anesthetic Techniques Used for Cesarean Delivery on Neonatal Cerebral and Renal Oxygenation
Brief Title: Cerebral and Renal Oxymetry and Anesthetic Techniques in Newborns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Antalya Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: AntalyaTRH 18
Record Dates: First submitted 2017-12-19; First posted 2018-01-03 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Cesarean Delivery Affecting Newborn
Keywords: Cesarean; newborn; cerebral and renal oxygenation; anesthesia
MeSH Terms: interventions — Spectroscopy, Near-Infrared; Anesthesia, Spinal; Anesthesia, General

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- spinal anesthesia (Active Comparator): Patients in this group were randomized to receive spinal anesthesia. (Near infrared spectroscopy (spinal anesthesia))
  Interventions: Device: Near infrared spectroscopy (spinal anesthesia)
- general anesthesia (Active Comparator): Patients in this group were randomized to receive general anesthesia. (Near infrared spectroscopy (general anesthesia)).
  Interventions: Device: Near infrared spectroscopy (general anesthesia)

INTERVENTIONS:
Device: Near infrared spectroscopy (spinal anesthesia) — effect of spinal anesthesia on regional renal and cerebral oxygen saturation in newborns
  Arms: spinal anesthesia
Device: Near infrared spectroscopy (general anesthesia) — effect of general anesthesia on regional renal and cerebral oxygen saturation in newborns
  Arms: general anesthesia

SUMMARY:
Neonatal adaptation to extrauterine life has many physiological changes in neonatal organ systems. These adaptative changes may be affected such as type of delivery and anesthesia management at birth. near infrared spectroscopy (NIRS) is a popular non-invasive method that can be used in newborns thus monitorize tissue oxygenation regularly. In this study we have purposed to compare the effects of general anesthesia versus spinal anesthesia on newborn's cerebral and renal oxygenation in elective cesarean operations

DETAILED DESCRIPTION:
The cases divided into two groups those spinal anesthesia group ( group:1; n:30 ) and general anesthesia group (group:2; n:30). The preoperative and intraoperative mean arterial pressures (MAP), heart rate (HR), arterial oxyhemoglobin saturation (SpO2), intraoperative blood loss values of pregnants and 1st-5th minute APGAR scores, preductal and postductal SpO2, perfusion index, heart rates, body temperature, cerebral and renal regional oxygen saturations of newborns after birth have been recorded.

ELIGIBILITY:
Inclusion Criteria:

* patients who undergo elective cesarean
* American Society of Anesthesiologists class 1 to 2
* Ability to consent
* Gestational age: from 37 to 41 weeks

Exclusion Criteria:

* Pulmonary disease
* History of allergic reaction to local anaesthetics
* Peripheral neuropathy
* Neurologic disease
* Coagulation disorders
* newborns with anomalies
* low birth weight newborns
* newborns needing neonatal resuscitation

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Change in renal and cerebral regional oxygenation (rSO2) in newborn | 60 minutes after birth
  Assessed at third and fifth minutes and then every 5 minutes after birth

SECONDARY OUTCOMES:
preductal SpO2 | 60 minutes after birth
  changes in preductal SpO2 after birth
postductal SpO2 | 60 minutes after birth
  changes in postductal SpO2 after birth
perfusion index | 60 minutes after birth
  changes in perfusion index after birth
body temperature | 60 minutes after birth
  changes in body temperature after birth
apgar scores | 1st and 5th minute after birth
  changes in apgar scores after birth

CONTACTS AND LOCATIONS:
Overall Officials: Ulku Arslan, MD, Study Director — Antalya Training and Research Hospital; Nilgun Kavrut Ozturk, MD, Principal Investigator — Antalya Training and Research Hospital; Ali Sait Kavakli, MD, Principal Investigator — Antalya Training and Research Hospital; Ozge Dagdelen, MD, Principal Investigator — Antalya Training and Research Hospital